CLINICAL TRIAL: NCT03640741
Title: Changes in Cerebral Oxygenation Studies Carried Out With the Use of Non-invasive Time-resolved Near-infrared Spectroscopy Device in Patients Undergoing Laparoscopy Procedure
Brief Title: Changes in Cerebral Oxygenation Studies During Laparoscopy Procedure
Status: Completed | Type: Observational
Sponsor: Nalecz Institute of Biocybernetics and Biomedical Engineering, Polish Academy of Sciences (Other)
Collaborators: Medical University of Lublin (Other)
Responsible Party: Sponsor
Other Study IDs: IAP_UMLub_GBox
Record Dates: First submitted 2018-07-17; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Increase in Intra-abdominal Pressure; Increase in Intracranial Pressure (ICP); Laparoscopy; Cerebral Perfusion and Oxygenation
Keywords: intra-abdominal pressure; intra-cerebral pressure; laparoscopy; brain perfusion; brain oxygenation; time-resolved near infrared spectroscopy
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Laparoscopy: The group consists of patients who undergoes laparoscopy procedure during which changes in cerebral oxygenation are estimated.
  Interventions: Procedure: Laparoscopy

INTERVENTIONS:
Procedure: Laparoscopy — The studies are carried out on patients who undergoes gynecological procedure that involves laparoscopy.

SUMMARY:
The motivation results from the fact, that an intra-abdominal pressure is correlated with cerebral perfusion, in a mechanism of reducing venous outflow. Moreover, elevated intra-abdominal pressure leads to increase in intracranial pressure and decrease of cerebral perfusion pressure.

The main aim of the study was to investigate an influence of increase in intra-abdominal pressure on cerebral oxygenation measured with the use of non-invasive optical technique.

DETAILED DESCRIPTION:
The investigators applied time resolved near infrared spectroscopy device in order to estimate changes in hemoglobin concentration in a brain during gynecological procedure that involves laparoscopy. The optodes were positioned on a forehead on left and right hemisphere.

The measurements were carried out during whole medical procedure, including anesthesia, start and stop of insufflation of abdominal cavity with carbon dioxide (CO2), surgical procedure, release of CO2 and waking up a patient. In those studies the special emphasis was put on a period of insufflation of abdominal cavity with CO2.

ELIGIBILITY:
Inclusion Criteria:

* laparoscopic procedure

Exclusion Criteria:

* no consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The studies are carried out on the gynecological ward of Medical University of Lublin what results in the fact that females were studied only.
Study Population: Patients of Gynecological Surgery Clinic
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2016-07-25 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
Distribution of time of flight of photons | 90 minutes (typically)
  Distribution of time of flight of photons measured at 2 wavelengths, 690 nm and 830 nm and at 2 spots on a forehead

SECONDARY OUTCOMES:
Cerebral oxygenation | 90 minutes (typically)
  Changes oxygenated (HbO2) and deoxygenated (Hb) hemoglobin concentrations expressed in micro Molars
Fluctuations of changes in Hb and HbO2 concentrations | 90 minutes (typically)
  Fourier transform of changes in concentrations of Hb and HbO2

CONTACTS AND LOCATIONS:
Overall Officials: Adam Liebert, Prof, Study Chair — Nalecz Institute of Biocybernetics and Biomedical Engineering

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bloomfield GL, Ridings PC, Blocher CR, Marmarou A, Sugerman HJ. Effects of increased intra-abdominal pressure upon intracranial and cerebral perfusion pressure before and after volume expansion. J Trauma. 1996 Jun;40(6):936-41; discussion 941-3. doi: 10.1097/00005373-199606000-00012. PMID 8656480
- [Background] Deeren DH, Dits H, Malbrain ML. Correlation between intra-abdominal and intracranial pressure in nontraumatic brain injury. Intensive Care Med. 2005 Nov;31(11):1577-81. doi: 10.1007/s00134-005-2802-2. Epub 2005 Sep 29. PMID 16193329
- [Background] Kacprzak M, Liebert A, Staszkiewicz W, Gabrusiewicz A, Sawosz P, Madycki G, Maniewski R. Application of a time-resolved optical brain imager for monitoring cerebral oxygenation during carotid surgery. J Biomed Opt. 2012 Jan;17(1):016002. doi: 10.1117/1.JBO.17.1.016002. PMID 22352652